CLINICAL TRIAL: NCT06222502
Title: Planning, Reminders and Micro-incentives to Increase Walking After Traumatic Brain Injury in Older Adults
Brief Title: Walking After Traumatic Brain Injury in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Timothy Morris (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Brandeis University (Other)
Responsible Party: Sponsor-Investigator, Timothy Morris, Principal Investigator, Northeastern University
Organization: Northeastern University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-06-23; P30AG048785 (NIH)
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury; TBI; Mild Traumatic Brain Injury; Moderate Traumatic Brain Injury
Keywords: Brain Injury; TBI; Walking; Exercise
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Brain Injuries; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Planning, Reminders, and Micro-Incentives (Experimental)
  Interventions: Other: Planning, Reminders, and Micro-Incentives
- Health Education (Active Comparator)
  Interventions: Other: Health Education

INTERVENTIONS:
Other: Planning, Reminders, and Micro-Incentives — Participants will schedule planned walks during weekly phone calls with study staff. Participants will receive reminders for planned walks and receive micro-incentives after completion.
  Arms: Planning, Reminders, and Micro-Incentives
Other: Health Education — Participants in this group will receive health education "tips" during weekly phone calls with study staff.
  Arms: Health Education

SUMMARY:
The purpose of this research is to learn if different behavioral interventions can change walking behaviors over 12-weeks, in older adults who have previously suffered a non-penetrating mild or moderate TBI.

Participants will provide information and be screened for eligibility via phone screening call (verification of age, confirmation that the participant is not currently on any medication that affects the central nervous system, and verification that the subject can participate in exercise, brief TBI history). Baseline testing will take place at the Center for Cognitive and Brain Health and Northeastern University Biomedical Imaging Center, for the baseline magnetic resonance imaging, in the interdisciplinary science and engineering complex on Northeastern University's campus. In person testing will take place over one session. The study period lasts 12 weeks, during which all participants will 1. Receive a weekly phone call with study staff and 2. Wear a wrist-worn Fit Bit tracker. A remote participation option is available for those who cannot travel to Northeastern University.

DETAILED DESCRIPTION:
Older adults are more affected by cognitive impairments due to TBI as compared to younger adults. In addition, older adults are at a much higher risk for sedentary behavior. To address this, we intend to test the effect of two behavioral interventions on walking participation of older adults with a history of mild or moderate TBI. Participants will be randomized to either the planning, reminders, and micro-incentives group or to the health education tips group which are delivered over the phone and available virtually. We will give each participant a Fit Bit for the duration of the study, and we will use it to track their walking. Our primary aim is to see if there is a difference in the activity levels between the groups. Our secondary aim is to see if the MRI data we collect shows intra-brain connections correlate with physical activity.

Our study is a 12-week two arm pilot randomized control trial-comparing two behavioral interventions. In one group, participants will have a weekly phone call with lab staff planning 5 days during each week that they plan on having a 30-minute walk. On the days of the walk, participants will receive either a text or an email, of their choice, reminding them of the planned walk. Participants will earn points for each planned walk completed; these can then be redeemed for a monetary reward at the end of the study. The other group will have a weekly phone call with lab staff where a health education tip is shared. Participants will also be provided a study FitBit where they will wear it during the times of the day when they are active.

Following recruitment and informed consent, each participant will come into ISEC for their baseline assessment. During this assessment they will fill out questionnaires on their health history to include: Physical Activity Readiness Questionnaire, Ohio state university TBI Questionnaire, PROMIS global health and NeuroQoL Questionnaires, Mediterranean diet adherence, International Physical Activity Questionnaire, Pittsburgh Sleep Quality Index, GAD-7, PHQ-9, BREQ-3 Physical Exercise Motivation, and the Physical Exercise Self Efficacy Questionnaire. Next, the participant will be asked to complete a battery of cognitive tests including: Digital and Paper Trail Making, Hopkins Verbal Learning Test, Letter and Category Fluency Test, and a mini mental status exam. This data will all be recorded via redcap. Next, the participant will undergo an MRI. This will take about an hour and the data will be uploaded to the Northeastern Cluster. Upon completion of the baseline session, each participant will be given a Fit Bit and assigned to the health education group or the planning, reminders, and micro-incentives group. Over the next 12 weeks, study staff will have access to the FitBit data collected and complete weekly calls with the participants, the content varying based on which group the participant is in. The final steps for the participants is their remote post testing where they will complete the same cognitive tasks and questionnaires as in their baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

• Suffered a mild or moderate traumatic brain injury within 3 months to 15 years prior to recruitment.

* TBI history will be assessed using the validated OSU TBI history questionnaire (Attachment 1). TBI severity will be defined as loss of consciousness of 0-30 minutes (mild) or >30 minutes and <24 hours (moderate). If no loss of consciousness was reported but post-traumatic amnesia was reported, then this is considered a mild TBI.

If clinical reports from the time of injury are available and Glasgow Coma Scale scores are available, then 13-15 is considered mild and 9-12 moderate. A clinical neurologist will review the de-identified OSU TBI forms for accuracy and confirm TBI severity.

* Men and women of all ethnicities/races and socio-economic status.
* 40-80 years.
* Signed Informed consent.
* Physically fit enough to undergo exercise as screened using the Physical Activity Readiness Questionnaire (PAR-Q) and the cardiovascular section of the Health History & Demographics Questionnaire. An affirmative response (i.e., "yes") to any single item regarding an individual's health status is grounds for the necessary medical clearance before enrollment.
* Normal or corrected-to-normal vision based on the minimal 20/20 standard in order to complete the cognitive tasks (below 20/20 vision).
* Able to speak, read, and write English.
* Ambulatory without pain or the assistance of walking devices.
* Reliable means of transportation (if participating in Boston).
* No diagnosis of a neurological disease.
* No intracerebral brain bleeds.
* Access to a mobile device, laptop or desktop computer with internet access and Bluetooth.

Exclusion Criteria:

* Diagnosis of a severe TBI (loss of consciousness >24 hours, post-traumatic amnesia > 7 days of a Glasgow Coma Scale of <9) or the presentation of skull breach.
* Prior diagnosis of cognitive or physical disability (severe asthma, epilepsy, chronic kidney disease, and dependence upon a wheelchair/walking aid).
* Not fluent in English.
* Undergoing any speech or physical therapy
* Not medically cleared for exercise.
* No history of vasovagal episodes (sudden drops in heart rate, poor perfusion, constant dizziness)
* History of intracerebral brain bleeds or strokes.
* Neurological condition (MS, Parkinson's, Dementia, MCI).
* Current treatment for congestive heart failure, angina, uncontrolled arrhythmia, DVT or other cardiovascular events.
* Myocardial infarction, coronary artery bypass grafting, angioplasty or other cardiac condition in the past year.
* Regular use of an assisted walking device.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Number of planned walks completed | 12 Weeks

SECONDARY OUTCOMES:
Functional connectivity of the anterior mid cingulate cortex, the dorsolateral and medial prefrontal cortex and diffusion metrics of the corpus callosum and association fiber tracts of the temporal and frontal lobes | 12 Weeks
Number of minutes walking per week and total number of steps per week | 12 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No